CLINICAL TRIAL: NCT04250948
Title: Perioperative Chemotherapy Plus PD-1 Antibody Compared With Perioperative Chemotherapy in the Locally Advanced Gastric Cancer: a Open-label, Phase 2 Randomised Controlled Trial
Brief Title: Efficacy of Perioperative Chemotherapy Plus PD-1 Antibody in the Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, President, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neoadjuvant PD-1/LAGC
Record Dates: First submitted 2019-11-10; First posted 2020-01-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer; Locally Advanced Solid Tumor
Keywords: Perioperative Therapy; PD-1 antibody; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — spartalizumab; Oxaliplatin; S 1 (combination); Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XELOX or SOX (Active Comparator): XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1
  Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Capecitabine: 1000mg/m2 Bid, d1-14, q3w;
  Neoadjuvant chemotherapy for 3 cycles, adjuvant chemotherapy for 5 cycles.
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Capecitabine
- JS001+XELOX or SOX (Experimental): XELOX: Oxaliplatin+Capecitabine; SOX: Oxaliplatin+S-1
  JS001: 240mg, ivdrip, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Capecitabine: 1000mg/m2 Bid, d1-14, q3w;
  Neoadjuvant chemotherapy for 3 cycles, adjuvant chemotherapy for 5 cycles.
  Interventions: Drug: JS001; Drug: Oxaliplatin; Drug: S1; Drug: Capecitabine

INTERVENTIONS:
Drug: JS001 — JS001, recombinant humanized anti-PD-1 monoclonal antibody for injection; 240mg ivdrip, d1, q3w.
  Other Names: PD-1 antibody
  Arms: JS001+XELOX or SOX
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2，iv drip for 2h，d1, q3w
Drug: S1 — S-1: 40~60mg Bid，d1~14, q3w
Drug: Capecitabine — Capecitabine: 1000mg/m2 Bid，d1-14, q3w
  Other Names: XELODA

SUMMARY:
For locally advanced gastric cancer (cT3-4aN+M0), neoadjuvant chemotherapy can downstage T and N stage, increase the resectability of tumor, and finally improve the long-term survival. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced gastric cancer could be a novel therapy to increase response rate and resectability and reduce recurrence rate. JS001 in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate tolerability, safety and efficacy of JS001 in combination with perioperative chemotherapy in locally advanced gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies in China with incidence and mortality both ranking the 2nd among malignancies in China. Surgery is the only possible way to cure gastric cancer, however, over 80-90% of gastric cancer patients in China are in advanced stage. Locally advanced gastric cancer (cT3-4aN+M0) could be cured by multi-disciplinary therapies including surgery, chemotherapy and radiotherapy. Neoadjuvant chemotherapy can downstage T and N stage, increase the resectability of tumor, and finally improve the long-term survival. However, the therapeutic effects remain unsatisfactory. PD-1 antibody has demonstrated its efficacy in metastatic gastric cancer and has been proved to be effective in neoadjuvant setting in lung cancer and melanoma. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced gastric cancer could be a novel therapy to increase response rate and resectability and reduce recurrence rate. JS001 in this study is a Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate tolerability, safety and efficacy of JS001 in combination with perioperative chemotherapy in locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent;
2. Histologically CT/MRI confirmed cT3-4aN+M0 gastric adenocarcinoma;
3. Consent to send tumor tissue from biopsy or resection for PD-L1, EBV, MSI detection;
4. Female or male, 18-75 years;
5. ECOG 0-1, no surgery contraindications;
6. Physical condition and adequate organ function to ensure the success of abdominal surgery;
7. Expected survival ≥3 months;
8. Adequate hematological, liver, renal and coagulation function;

1) Platelet (PLT) count ≥100,000 /mm3; 2) Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6) Glycosylated hemoglobin (HbA1c) <7.5%; 7) Total bilirubin (TBIL) level ≤1.5×ULN; 8) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 9) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 10) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min; 11) Thyroid stimulating hormone (TSH) ≤ULN; 12) Normal serum free thyroid hormone (T4); 13) Normal serum free triiodothyronine (T3); 14) Serum amylase ≤1.5×ULN; 15) Lipase ≤1.5×ULN.

9.Females of child bearing age must have a negative pregnancy test, and have to take contraception measures and avoid breast feeding during the study and for 3 months after the last dose; male subjects must agree to taken contraception measures during the study and for 3 months after the last dose.

Exclusion Criteria:

1. Known allergy to study drug or excipients, or allergy to similar drugs;
2. Patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured localized tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ;
3. Uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment;
4. Weight loss >20% within 2 weeks before recruitment;
5. Unable to swallow study drug;
6. Prior chemotherapy, radiotherapy, surgery for gastric cancer;
7. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent;
8. Prior therapy with tyrosine kinase inhibitor within 2 weeks.
9. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy;
10. Have vaccination with attenuated live vaccines within 4 weeks prior to initiation of the study treatment or plan to vaccinate during the study;
11. Poorly controlled hypertension or diabetes;
12. With bleeding tendency, or evident hemoptysis or other hemorrhagic events (e.g. gastrointestinal hemorrhage, hemorrhagic gastric ulcer) within 2 months prior to initiation of study treatment, or presence of hereditary or acquired bleeding or thrombotic tendency (e.g. hemophilia, coagulopathy, thrombocytopenia, etc.), or current/long-term thrombolytic or anticoagulant therapy (except aspirin ≤100 mg/day);
13. Present or history of any autoimmune disease;
14. With active tuberculosis or receiving previous anti-tuberculosis therapy within one year;
15. Diagnosed with interstitial pneumonia, non-infectious pneumonia, pulmonary fibrosis, acute lung disease;
16. Pregnancy or breast feeding;
17. Human immunodeficiency virus (HIV) infection (HIV antibody positive), or active hepatitis C virus (HCV) infection (HCV antibody positive), or active hepatitis B virus (HBV) infection (HBsAg or HBcAb positive, and HBV-DNA ≥2000 IU/ml (copies/ml)), or other severe infection requiring systemic antibiotic treatment, or unexplained body temperature >38.5℃ during screening period/before study treatment;
18. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
TRG0/1 | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Pathological tumor regression grade 0/1

SECONDARY OUTCOMES:
pCR | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Pathological complete response
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
Recurrence free survival (RFS) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented recurrence
Objective response rate (ORR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Defined as the proportion of patients whose tumors shrink for a certain period of time
Disease control rate (DCR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years]
  Defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time
Overall survival (OS) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan SQ, Nie RC, Jin Y, Liang CC, Li YF, Jian R, Sun XW, Chen YB, Guan WL, Wang ZX, Qiu HB, Wang W, Chen S, Zhang DS, Ling YH, Xi SY, Cai MY, Huang CY, Yang QX, Liu ZM, Guan YX, Chen YM, Li JB, Tang XW, Peng JS, Zhou ZW, Xu RH, Wang F. Perioperative toripalimab and chemotherapy in locally advanced gastric or gastro-esophageal junction cancer: a randomized phase 2 trial. Nat Med. 2024 Feb;30(2):552-559. doi: 10.1038/s41591-023-02721-w. Epub 2024 Jan 2. PMID 38167937